CLINICAL TRIAL: NCT00330395
Title: A Multicenter, Sequential-Panel, Open-Label, Noncomparative Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Caspofungin Acetate in Neonates and Infants Less Than 3 Months of Age.
Brief Title: Open, Pharmacokinetic Study of Caspofungin in Neonates and Infants (0991-058)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0991-058; MK0991-058; 2006_025
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Candidiasis
MeSH Terms: conditions — Candidiasis | interventions — Caspofungin

INTERVENTIONS:
Drug: caspofungin acetate — Duration of Treatment 28 Days
  Other Names: MK0991

SUMMARY:
The purpose of this study is to test the amount of caspofungin found in the blood of neonate and infants <3 months of age following treatment with caspofungin at 25 mg/m2. Another purpose is to test the safety of caspofungin in treating neonates and infants with Candida infections (a certain type of fungal infection).

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants <3 months of age
* Patient has a body weight greater than or equal to 500 grams
* Patient has documented or highly suspected Candida infection

Exclusion Criteria:

* Patient is greater than 3 months of age
* Patient has a body weight of less than 500 grams
* Patient does not meet certain laboratory testing criteria
* Patient is hemodynamically unstable, exhibits hemodynamic compromise or is not expected to survive at least 5 days
* Patient has documented HIV infection of any stage
* Patient has a history of allergy, hypersensitivity, or serious reaction to caspofungin or another member of the echinocandin class

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2006-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of drug exposure

SECONDARY OUTCOMES:
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Saez-Llorens X, Macias M, Maiya P, Pineros J, Jafri HS, Chatterjee A, Ruiz G, Raghavan J, Bradshaw SK, Kartsonis NA, Sun P, Strohmaier KM, Fallon M, Bi S, Stone JA, Chow JW. Pharmacokinetics and safety of caspofungin in neonates and infants less than 3 months of age. Antimicrob Agents Chemother. 2009 Mar;53(3):869-75. doi: 10.1128/AAC.00868-08. Epub 2008 Dec 15. PMID 19075070
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html